CLINICAL TRIAL: NCT03934580
Title: Postprandial Effects of a Hallucinatory Meal on Appetite Regulation: a Randomized Cross-over Pilot Trial
Brief Title: Postprandial Effects of a Hallucinatory Meal on Appetite Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 183121
Record Dates: First submitted 2019-04-23; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Change in Subjective Appetite Score (VAS)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hallucinated meal (Experimental): A breakfast meal (white bread plus ham and cheese with 250 ml still water) is hallucinated under hypnosis by participants for 15 minutes
  Interventions: Other: hallucinated meal
- real meal (Active Comparator): A real meal (white bread plus ham and cheese with 250 ml still water) is consumed by participants in 15 minutes
  Interventions: Other: Real meal

INTERVENTIONS:
Other: hallucinated meal — a breakfast meal (white bread plus ham and cheese with 250 ml still water) is hallucinated by participants under hypnosis
  Arms: hallucinated meal
Other: Real meal — A real breakfast (white bread plus ham and cheese with 250 ml still water) is consumed by participants
  Arms: real meal

SUMMARY:
Several and complex mechanisms are involved in the regulation of appetite and food intake in humans. By means of rapid hypnosis techniques, it is possible to induce some individuals to hallucinate a meal.

The same meal (breakfast) is administered as i) a real meal and ii) is evoked as a hallucination under hypnosis in healthy postmenopausal women. The aim of this pilot randomized-controlled cross-over trial is to assess appetite sensation and the blood levels of the appetite-related hormones in the participants.

DETAILED DESCRIPTION:
The regulation of appetite is crucial to control food intake and consequently body weight. Hypnosis has been successfully used to modulate gastrointestinal functions, by imagining eating food.

In the present pilot trial, the investigators search to investigate the effects a hallucinatory meal by hypnosis on subjective appetite and appetite hormone blood levels. Hence, two different breakfast meals are randomly administered to eight healthy postmenopausal women, in a crossover design, consisting of i) a hallucinatory breakfast meal (HB) and ii) a real breakfast meal (RB). On each test day, participants undergo baseline measurements, including appetite sensation and blood sample, then the test meal is hallucinated or served. Subjective appetite is assessed each 30 minutes for 4 hours and half, while blood samples are taken at 20', 60', 90' and 180 minutes. At the end of each session, participants are instructed to fill in a food record for the following 3-days.

ELIGIBILITY:
Inclusion Criteria:

* female gender,
* ability to develop a visual hallucination during hypnosis,
* body mass index (BMI) range 20-27 kg/m2,
* menopausal status

Exclusion Criteria:

* smoking,
* breakfast skipping,
* current intake of any supplements,
* current use of any drug,
* presence of any pathological conditions, including mental and eating disorders,
* any alimentary restrictions or specific diets,
* allergies or food intolerances or dislikes of the offered breakfast-meal,
* being a shift or night workers,
* unable to give a written informed consent

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in subjective appetite score (VAS) | 270 minutes
  changes in subjective appetite score as measured by VAS after the hallucinated meal compared to the changes in subjective appetite score after the real meal

SECONDARY OUTCOMES:
Changes in circulating concentrations of PYY | 180 minutes
  changes in circulating concentrations of PYY after the hallucinated meal compared to the changes after the real meal
Changes in circulating concentrations of GLP-1 | 180 minutes
  changes in circulating concentrations of GLP-1 after the hallucinated meal compared to the changes after the real meal
Changes in circulating concentrations of ghrelin | 180 minutes
  changes in circulating concentrations of ghrelin after the hallucinated meal compared to the changes after the real meal
Changes in circulating concentrations of NPY | 180 minutes
  changes in circulating concentrations of NPY after the hallucinated meal compared to the changes after the real meal
Changes in circulating concentrations of orexin-A | 180 minutes
  changes in circulating concentrations of orexin-A after the hallucinated meal compared to the changes after the real meal
Changes in circulating concentrations of leptin | 180 minutes
  changes in circulating concentrations of leptin after the hallucinated meal compared to the changes after the real meal
Changes in circulating concentrations of alpha-MSH | 180 minutes
  changes in circulating concentrations of alpha-MSH after the hallucinated meal compared to the changes after the real meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, AT, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cioffi I, Gambino R, Rosato R, Properzi B, Regaldo G, Ponzo V, Pellegrini M, Contaldo F, Pasanisi F, Ghigo E, Bo S. Acute assessment of subjective appetite and implicated hormones after a hypnosis-induced hallucinated meal: a randomized cross-over pilot trial. Rev Endocr Metab Disord. 2020 Sep;21(3):411-420. doi: 10.1007/s11154-020-09559-4. PMID 32418064